CLINICAL TRIAL: NCT04959630
Title: Effectiveness of an Immersive Virtual Reality Environment on Curricular Training for Complex Cognitive Skills in Liver Surgery: A Multicentric Crossover Randomized Trial
Brief Title: Immersive Virtual Reality Environment for Complex Cognitive Skills Curricular Training in Liver Surgery
Acronym: LiVeRTrainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, GIHeelkunde, Department of GI Surgery, University Hospital, Ghent
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: B6702020000275
Record Dates: First submitted 2021-06-21; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Hepatobiliary Neoplasm
Keywords: surgical education; 3D reconstruction; virtual reality; surgical planning; cognitive knowledge training; decision making
MeSH Terms: interventions — Environment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Group A received first five patient cases and 3D models via DI and another five cases in the VR environment
  Interventions: Behavioral: Clinical decision making based on visualizing liver 3D models in Virtual Reality (VR) environment or via a Desktop Interface (DI)
- Group B (Other): Group B received first five patient cases and 3D models via VR and another five cases in the DI.
  Interventions: Behavioral: Clinical decision making based on visualizing liver 3D models in Virtual Reality (VR) environment or via a Desktop Interface (DI)

INTERVENTIONS:
Behavioral: Clinical decision making based on visualizing liver 3D models in Virtual Reality (VR) environment or via a Desktop Interface (DI) — Visualizing 3D models of livers for preoperative surgical planning via two different environment: DI and VR in sequential order

SUMMARY:
Investigators hypothesize that a virtual reality (VR) environment enhances general surgery residents' performance compared to Desktop Interface (DI)-based visualization of 3D models in decision making for patients with liver tumors. To determine this, a proficiency-based stepwise training curriculum for preoperative planning has been developed using both modalities. The overall objective of the curriculum is that by the end of the training program, residents would be able to formulate a treatment plan for patients with liver tumors.

ELIGIBILITY:
Inclusion Criteria:

• General surgery residents irrespective of their postgraduate year

Exclusion Criteria:

* No inform consent
* Residents of other specialties

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Residents' decision-making accuracy | Immediately after completing the educational intervention
  Residents' decision-making accuracy when reviewing patient data and 3D liver models using DI or VR, measured by comparing their performance to experts' opinions.
  The measurement tool will be a questionnaire consisting of ten questions, rate of correct answers will be recorded (e.g. 8/10 correct answers) and higher scores mean a better outcome.
  Minimum score=0; Maximum score=10.

SECONDARY OUTCOMES:
Cognitive knowledge retention | Baseline and immediately after completing the educational intervention
  Retention of knowledge assessed by validated multiple choice questions. Questionnaire consisted of 15 questions will be used, rate of correct answers will be recorded (e.g. 8/15 correct answers), and higher scores mean a better outcome.
  Minimum score=0; Maximum score=15.
Residents' scores in recognizing intrahepatic structures and liver segments | Immediately after completing the educational intervention
  Assessed by recognizing intrahepatic structures and 8 liver segments. Questionnaire consisted of 22 questions will be used, rate of correct answers will be recorded (e.g. 8/22 correct answers), and higher scores mean a better outcome.
  Minimum score=0; Maximum score=22.
Time needed to devise a surgical plan using the DI or VR platform | Immediately after completing the educational intervention
  Assessed by total time needed to make decision for 10 patient cases in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wouter Willaert, MD, PhD, Principal Investigator — University Hospital, Ghent; Roberto Troisi, MD, PhD, Principal Investigator — Federico II University
Locations (2):
- Ghent University Hospital, Ghent, Belgium
- Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD are to be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication

REFERENCES:
- [Derived] Rashidian N, Giglio MC, Van Herzeele I, Smeets P, Morise Z, Alseidi A, Troisi RI, Willaert W. Effectiveness of an immersive virtual reality environment on curricular training for complex cognitive skills in liver surgery: a multicentric crossover randomized trial. HPB (Oxford). 2022 Dec;24(12):2086-2095. doi: 10.1016/j.hpb.2022.07.009. Epub 2022 Jul 21. PMID 35961933

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04959630/Prot_SAP_000.pdf